CLINICAL TRIAL: NCT01877629
Title: A Single-center, Open-label, Two-period, Two-treatment, Crossover, Single-dose Study in Healthy Female and Male Subjects to Assess the Pharmacokinetics, Safety, and Tolerability of Two Different Formulations of ACT-129968
Brief Title: Clinical Study to Assess the Pharmacokinetics, Safety, and Tolerability of ACT-129968 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AC-060-104
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Tolerability; Safety; ACT-129968
MeSH Terms: interventions — 2-(2-(1-naphthoyl)-8-fluoro-3,4-dihydro-1H-pyrido(4,3-b)indol-5(2H)-yl)acetic acid; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT-129968 tablet/capsules (Experimental): Subjects attend two treatment periods. In the first treatment period subjects receive a single, oral dose of ACT-129968 500 mg administered as a tablet (1 tablet, 500 mg) in the fasted state. In the second treatment period subjects receive a single, oral dose of ACT-129968 500 mg administered as capsules (2 capsules, 250 mg each) in the fasted state. There is a 7-9 day washout period between the first treatment period and the second treatment period.
  Interventions: Drug: ACT-129968 500 mg tablet; Drug: ACT-129968 250 mg capsule
- ACT-129968 capsules/tablet (Experimental): Subjects attend two treatment periods. In the first treatment period subjects receive a single, oral dose of ACT-129968 500 mg administered as capsules (2 capsules, 250 mg each) in the fasted state. In the second treatment period subjects receive a single, oral dose of ACT-129968 500 mg administered as a tablet (1 tablet, 500 mg each) in the fasted state. There is a 7-9 day washout period between the first treatment period and the second treatment period.
  Interventions: Drug: ACT-129968 500 mg tablet; Drug: ACT-129968 250 mg capsule

INTERVENTIONS:
Drug: ACT-129968 500 mg tablet — ACT-129968, a tetrahydropyridoindole derivative, is a chemoattractant receptor homologous molecule expressed on T helper 2 cells (CRTH2) antagonist
Drug: ACT-129968 250 mg capsule — ACT-129968, a tetrahydropyridoindole derivative, is a chemoattractant receptor homologous molecule expressed on T helper 2 cells (CRTH2) antagonist

SUMMARY:
To explore the pharmacokinetics (PK) of a single dose of two different formulations of ACT-129968, i.e., tablet versus capsule and to evaluate the safety and tolerability of a single dose of two different formulations of ACT-129968, i.e., tablet versus capsule.

DETAILED DESCRIPTION:
A total of 10 female and 10 male healthy subjects will be enrolled and will attend two treatment periods, separated by a 7-9 day washout. Over these two periods, two formulations of ACT-129968 (Treatment A: two capsules, 250 mg each; Treatment B: one tablet, 500 mg) will be administered in the sequence A/B or B/A to 10 subjects (5 females and 5 males) per sequence as determined by randomization.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure.
* Women must have

  * a negative serum pregnancy test at screening and
  * a negative urine pregnancy test pre-dose on Day-1 of each treatment period.
* Women of childbearing potential must consistently and correctly use (from screening, during the entire study, and for at least 28 days after last study drug intake) a reliable method of contraception with a failure rate of < 1% per year, be sexually inactive, or have a vasectomized partner.

Women not of childbearing potential are defined as post-menopausal (i.e., spontaneous amenorrhea for at least 1 year without an alternative medical cause) or surgically or naturally sterile.

* No clinically significant findings on the physical examination at screening.
* Body mass index (BMI) of 18.0 to 28.0 kg/m^2 (inclusive) at screening.
* Systolic blood pressure (SBP) 100-145 mmHg, diastolic blood pressure (DBP) 50-90 mmHg, and pulse rate (PR) 45-90 bpm (inclusive), measured on the dominant arm (dominant arm = writing arm) after 5 minutes in the supine position at screening.
* 12-lead electrocardiogram (ECG) without clinically relevant abnormalities, measured after 5 minutes in the supine position at screening.
* Hematology, clinical chemistry, and urinalysis test results not deviating from the normal range to a clinically relevant extent at screening.
* Negative results from urine drug screen and breath alcohol test at screening and on admission to the unit (Day-1) in Period 1 and Period 2.
* Ability to communicate well with the investigator, in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Pregnant or lactating women.
* Known allergic reactions or hypersensitivity to any excipient of the drug formulation(s).
* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism, or excretion of the study drug (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* History or clinical evidence of allergic rhinitis or asthma.
* Veins unsuitable for intravenous puncture on either arm (e.g., veins that are difficult to locate, access, or puncture, veins with a tendency to rupture during or after puncture).
* Previous exposure to the study medication.
* Treatment with another investigational drug within 3 months prior to screening or participation in more than four investigational drug studies within 1 year prior to screening.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* Excessive caffeine consumption, defined as 800 mg per day at screening.
* Alcohol consumption of > 21 units/week or > 3 units/day.
* Smoking within 3 months prior to screening.
* Previous treatment with any prescribed or over-the-counter medications (including herbal medicines such as St John's Wort) within 2 weeks prior to first study drug administration.
* Loss of 250 mL or more of blood within 3 months prior to screening.
* Positive results from the hepatitis serology (Hepatitis B surface antigen and anti-hepatitis C virus), except for vaccinated subjects or subjects with past but resolved hepatitis (defined as positive finding for antibodies but negative findings for antigens), at screening.
* Positive results from the human immunodeficiency virus serology at screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Legal incapacity or limited legal capacity at screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07-01; Primary Completion 2011-07-01 (Actual); Study Completion 2011-07-01 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration-time curve from time zero to time t of the last measured concentration above the limit of quantification (AUC0-t). | Up to 48 h in each treatment period (1 and 2)
  The plasma PK parameters for ACT-129968 will be derived by non-compartmental analysis of the plasma concentrationtime profiles.
The area under the plasma concentration-time curve from zero to infinity (AUC0-infinity). | Up to 48 h in each treatment period (1 and 2)
  The plasma PK parameters for ACT-129968 will be derived by non-compartmental analysis of the plasma concentrationtime profiles.
The maximum plasma concentration (Cmax) | Up to 48 h in each treatment period (1 and 2)
  The plasma PK parameters for ACT-129968 will be derived by non-compartmental analysis of the plasma concentrationtime profiles.
The time to reach maximum plasma concentration (tmax) | Up to 48 h in each treatment period (1 and 2)
  The plasma PK parameters for ACT-129968 will be derived by non-compartmental analysis of the plasma concentrationtime profiles.
The terminal elimination half-life (t½) | Up to 48 h in each treatment period (1 and 2)
  The plasma PK parameters for ACT-129968 will be derived by non-compartmental analysis of the plasma concentrationtime profiles.

SECONDARY OUTCOMES:
Change from baseline to each time point of measurement during each treatment period and to EOS in supine blood pressure | Up to 13 days
  mmHg
Change from baseline to each time point of measurement during each treatment period and to EOS in pulse rate | Up to 13 days
  bpm
Body weight at baseline and end of study visit | Up to 13 days
Change from baseline to EOS for hematology | Up to 13 days
Change from baseline to EOS for clinical chemistry | Up to 13 days
Change from baseline to EOS for pregnancy serum test | Up to 13 days
Change from baseline to EOS for virus serology | Up to 13 days
Change from baseline to each time point of measurement during each treatment period and to EOS in ECG variables | Up to 13 days
  ECG variables are to be recorded at rest using a standard 12-lead ECG
Number of patients with treatment-emergent ECG abnormalities for each treatment period | from study drug administration on Day 1 up to 48 hours post-dose
Number of patients with treatment-emergent physical examination abnormalities at EOS | Up to 13 days
Number of patients with treatment-emergent AEs and SAEs for each treatment period | from study drug administration on Day 1 up to 48 hours post-dose
Number of patients with AEs leading to premature discontinuation of study drug | Entire duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Baldoni, PharmD, PhD, Study Director — Actelion
Locations (1):
- PHAROS GmbH Clinical Research, Ulm, Germany

REFERENCES:
- [Derived] Baldoni D, Mackie A, Gutierrez M, Theodor R, Dingemanse J. Setipiprant, a selective oral antagonist of human CRTH2: relative bioavailability of a capsule and a tablet formulation in healthy female and male subjects. Clin Ther. 2013 Nov;35(11):1842-8. doi: 10.1016/j.clinthera.2013.09.003. Epub 2013 Oct 4. PMID 24095247